CLINICAL TRIAL: NCT01310751
Title: Randomized Double-blind Study of Inhaled Iloprost for the Treatment of Pulmonary Hypertension (PH) and Pulmonary Hypertensive Crisis (PHC) After Repair of Congenital Heart Disease (CHD)
Brief Title: Study of Inhaled Iloprost in Pediatric Pulmonary Hypertension (PH) After Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhuoming, chief cadiologist,Director of ICU, Cardiac intensive Care Unit,Department of Thoracic and Cardiovascular Sugery,Shanghai Children's Medical Center., Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SJTUMS-200903
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iloprost nebuliser solusion (Experimental): 50 ng/kg/min
  Interventions: Drug: iloprost nebuliser solusion
- distilled water (Placebo Comparator): 2ml
  Interventions: Drug: distilled water

INTERVENTIONS:
Drug: iloprost nebuliser solusion — 50 ng/kg/min inhalation for 10 minutes, q2h for 2 days
  Other Names: Venatvis
  Arms: iloprost nebuliser solusion
Drug: distilled water — 2 ml per session
  Other Names: placebo
  Arms: distilled water

SUMMARY:
The aim of this study is to determine whether inhaled iloprost can be used to prevent and treat PH and PHC while in children after operation of CHD

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a significant contributor to the postoperative morbidity and mortality of congenital heart disease. Inhaled iloprost has been approved for the treatment of adults with PH, but little is known about the effects in children with PH.

Iloprost is a prostacyclin analogue. When applied by inhalation, it selectively dilates pulmonary vessels without side affecting the systemic circulation. There is no RCTs of iloprost have previously been performed in this indication.

ELIGIBILITY:
Inclusion Criteria:

Before corrective procedure for CHD, two of bellow ten criteria should be met

1. Pulse SaO2 smaller than 93% in left-right shunt CHD case (in room air)
2. EKG: right ventricular hypertrophy, right atrial dilatation
3. Chest X-ray: enhanced vascular signs in trans-hilar, loss of blood vessal in bilateral lung fields, pulmonary arterial trunk dilatation, right ventricular enlargement
4. Cardiac echocardiography: fast tricuspid or pulmonary valve regurgitant velocity, ventricular and aortic level bidirectional shunt, or even right-to-left shunt
5. Under-filling of pulmonary capillary, 'pruning' of the peripheral blood vessels
6. Pp/Ps greater than 0.75
7. Qp/Qs smaller than 1.5
8. PVR grater than 9 Wood Unit/m2
9. Rp/Rs graeter than 0.5

Exclusion Criteria:

After corrective procedure for CHD:

1. Deficient anatomy associated with remained intracardiac shunts and severe artrio-ventricular regurgitation
2. Severe arrhythmia led to low cardiac output
3. PLT smaller than 50,000*109/L and obvious bleeding

Ages: 9 Days to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary end point is a composite variable (incidence rate of any events) consisting of reactive PH, PHC and death requiring additional pharmacological or other support administered within the first 48 hours after receiving study drug. | The pulmonary heamodynamic variable is measured before, after ilkoprost inhalation instantly and 30-min later.
  Reactive PH is defined as Pp/Ps greater than 0.5 for more than 30min.
  End point of observation: in case of Pp/Ps greater than 0.5 for more than 30min or Pp/Ps greater than 1 for any time period, drug inhalation will be immediately stopped and other therapies such as NO inhalation and/or iloprost 80 ng/kg/min inhalation will be resorted to treat pulmonary hypertension.

SECONDARY OUTCOMES:
Change from base line of pulmonary heamodynamic measurements: Pp/Ps, PVRI, SVRI | The heamodynamic variable is measured before, after iloprost inhalation instantly and 30-min later.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhuo-ming, M.D., PhD., Study Director — Cardiac intensive Care Unit,Department of Thoracic and Cardiovascular Sugery,Shanghai Children's Medical Center
Locations (1):
- Cardiac intensive Care Unit,Department of Thoracic and Cardiovascular Sugery,Shanghai Children's Medical Center, Shanghai, China